CLINICAL TRIAL: NCT00626145
Title: Long Term Functional Evaluation After Intracoronary Delivery of Autologous Bone Marrow Mononuclear Cells in Patients With ST-Elevation Myocardial Infarction
Brief Title: Long Term Follow-up of Autologous Bone Marrow Mononuclear Cells Therapy in STEMI
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Haichang Wang / Director of Department of Cardiology of Xijing Hospital, Xijing Hospital of Fourth Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00200301
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Last update posted 2008-02-29 (Estimated); Status verified 2008-02

CONDITIONS: Myocardial Infarction
Keywords: BMMNC; STEMI; stem cell; intracoronary delivery
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Patients receive intracoronary injections of saline 7 days after PCI.
  Interventions: Procedure: saline infusion
- 2 (Experimental): Patients receive intracoronary injections of autologous bone marrow mononuclear cells 7 days after PCI.
  Interventions: Procedure: autologous bone marrow mononuclear cells infusion

INTERVENTIONS:
Procedure: saline infusion — Patients receive intracoronary injections of saline 7 days after PCI.
  Other Names: saline placebo; placebo control
  Arms: 1
Procedure: autologous bone marrow mononuclear cells infusion — Patients receive intracoronary injections of autologous bone marrow mononuclear cells 7 days after PCI.
  Other Names: autologous BMMC infusion; autologous bone marrow mononuclear cells transplantation; autologous BMMC intracoronary injection
  Arms: 2

SUMMARY:
The benefit of current reperfusion therapies for ST-elevation myocardial infarction (STEMI) is limited by post-infarction left ventricular (LV) dysfunction. Many clinic trails showed the short term outcome of bone marrow stem cell transplantation for MI patients, but rare report of long term follow-up results. Our aim was to investigate 4 years' efficacy and LV functional improvement of autologous bone marrow mononuclear cells (BMMC) transplantation in patients with ST-elevation myocardial infarction.

DETAILED DESCRIPTION:
The benefit of current reperfusion therapies for ST-elevation myocardial infarction (STEMI) is limited by post-infarction left ventricular (LV) dysfunction. Many clinic trails showed the short term outcome of bone marrow stem cell transplantation for MI patients, but rare report of long term follow-up results.

Aim is to evaluate the long term efficiency of unselected bone marrow mononuclear cells in treatment of patients with ST-elevation myocardial infarction (STEMI), especially with regard to the left ventricular function. The cells are delivered by intracoronary infusion 7 days after the PCI. Outcomes including LVEF, myocardial viability and coronary artery status are assessed by echocardiography, SPECT and coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* ST segment elevation myocardial infarction, according to the WHO definition.
* <24 hour from the origin of symptoms.
* Single left anterior descending coronary artery disease.
* Successful revascularization of culprit lesion with PCI.
* Age between 45 and 65 years old.
* Written informed consent.

Exclusion Criteria:

* Previous MI.
* Cardiomyopathy.
* Atrial fibrillation or fluctuation.
* Previous heart surgery.
* Severe valvular heart disease.
* Disease of the hematopoetic system.
* NYHA functional class IV at baseline.
* Severe renal, lung and liver disease or cancer.
* Significant coronary lesion in one or more major coronary vessels, requiring revascularization.
* Intra-cardiac thrombus.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2003-03; Primary Completion 2008-03 (Estimated); Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular Ejection Fraction(LVEF) | 1, 3, 6 months, 1, 4 years

SECONDARY OUTCOMES:
in-stent restenosis | 1, 3, 6 months, 1, 4 years
cardiac shock | 1, 3, 6 months, 1, 4 years
myocardial viability of the infarcted area | 1, 3, 6 months, 1, 4 years
end-diastolic Volume/end-systolic Volume(EDV/ESV) | 1, 3, 6 months, 1, 4 years
wall motion score index(WMSI) | 1, 3, 6 months, 1, 4 years
cumulative MACE(including cardiac death, non-fetal myocardial infarction and target lesion revascularization) | 1, 3, 6 months, 1, 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Haichang Wang, MD,PHD, Principal Investigator — Xijing Hospital
Locations (1):
- Department of Cardiology in Xijing Hospital, Xi'an, Shaanxi, China